CLINICAL TRIAL: NCT01874834
Title: Cardiopulmonary Responses to Exposure to Ozone and Diesel Exhaust With Moderate Exercise in Healthy Adults
Brief Title: Cardiopulmonary Responses to Exposure to Ozone and Diesel Exhaust
Acronym: DEPOZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Environmental Protection Agency (EPA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Madden, Research Biologist, Environmental Protection Agency (EPA)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Diagnostic
Other Study IDs: EPA 09-1344
Record Dates: First submitted 2013-06-07; First posted 2013-06-11 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Respiratory Depression; Blood Pressure
Keywords: ozone; diesel; lung function; cardiac electrophysiology; mediators of inflammation and clotting
MeSH Terms: conditions — Respiratory Insufficiency; Thrombosis | interventions — Ozone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Filtered air exposure (Placebo Comparator): 2 hr exposure to clean, filtered air with intermittent exercise
  Interventions: Other: ozone
- Ozone (Experimental): 2 hr exposure to 300 ppb ozone with intermittent exercise
  Interventions: Other: ozone
- Diesel Exhaust, No ozone (Experimental): 2 hr exposure to whole diesel exhaust (300 ug/m3; gases + particles) with intermittent exercise; no ozone
  Interventions: Other: ozone
- Ozone + Diesel Exhaust (Experimental): 2 hr exposure to a combination of 300 ppb ozone an 300 ug/m3 whole diesel exhaust with intermittent exercise
  Interventions: Other: ozone

INTERVENTIONS:
Other: ozone — Exposure to 300 ppb ozone with intermittent exercise about 20 hr after exposure to each arm (ie, either air, ozone, diesel exhaust, or ozone combined with diesel exhaust)
  Other Names: cas # 10028-15-6; trioxygen

SUMMARY:
The US EPA Clean Air Multiyear research program is moving toward a multi-pollutant approach to the assessment of air pollution in response to recommendations by the NRC 2004 and the BOSC in 2005. Such an approach better reflects the complexity of real-world air pollution problems and parallels evolving scientific and regulatory considerations. Ozone (O3) and diesel exhaust (DE) generally are major and important components of ambient air pollution. This proposed study will address the agency's goals by investigating the cardiopulmonary health effects in healthy human subjects co-exposed to O3 and DE. The findings derived from these exposures will provide NCEA findings for risk assessments of O3 and DE, as well as the Office of Air and Radiation (includes OTAQ and OAQPS) with information relevant to possible modulation of PM-induced health effects and responses by a gaseous co-pollutant for potential standard setting. Additionally the findings will address the fundamental driving principle of the Clean Air Research strategy related to reduction of health due to air pollutant exposures.

DETAILED DESCRIPTION:
Numerous epidemiological studies have demonstrated an association between acute and chronic exposure to air pollution and various adverse cardiopulmonary effects including mortality, respiratory tract infections, exacerbation of asthma symptoms, chronic bronchitis, ischemic heart disease, and stroke [1] and other health effects. Understanding the components responsible for these effects is difficult because ambient air pollution is a complex mixture of gases and particulate matter (PM). In this complex mixture of ambient air pollution, ozone (O3) and diesel exhaust (DE) are generally major and important components. Controlled exposure of volunteers to either pollutant have resulted in biological effects such as lung physiological changes. However it is not known if co-exposure to both pollutants, similar to polluted ambient air, can induce additive or synergistic effects. Additionally it is also uncertain if exposure to DE, or DE with O3, can alter a subsequent exposure to O3 similar to multiple day exposures that the general population receives. This study proposes to examine whether co-exposures to O3 and DE can induce additive or synergistic effects, and whether a previous DE exposure alters a response upon subsequent exposure to O3. The potential effects of O3 on cardiac electrophysiology are also not clear.

Approximately 15 healthy non-smoking volunteers between the ages of 18 and 55 will be exposed in a controlled manner to O3 (approximately mean concentration of 0.3 ppm over the 2 hr exposure period), or diesel exhaust (DE; ~300 µg/m3), or a combined O3 and DE exposure while undergoing moderate intermittent exercise at the EPA Human Studies Facility. A clean air exposure will serve as a control. Primary endpoints for evaluating health effects and surrogate responses are changes in lung function and heart rate variability. In addition, other cardiopulmonary and vascular biological endpoints will be measured, as well as markers of exposure and genetic markers of susceptibility.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women between 18 and 55 years of age
* Physical conditioning allowing intermittent, moderate exercise for 2 hours
* Normal lung function:

  1. FVC > 75 % of that predicted for gender, ethnicity, age and height.
  2. FEV1 > 75 % of that predicted for gender, ethnicity, age and height.
  3. FEV1/FVC ratio > 75 % of predicted values.
* Oxygen saturation > 96 %.

Exclusion Criteria:

* A history of acute and chronic cardiovascular disease, chronic respiratory disease, diabetes, rheumatologic diseases, immunodeficiency state, and acute respiratory illness within 4 weeks.
* Subjects who are asthmatic or have a history of asthma.
* Allergic to chemical vapors or gases.
* Any allergic symptoms during the time of participation in the study
* Female subjects who are currently pregnant, attempting to become pregnant, or breastfeeding
* Subjects unwilling or unable to stop taking vitamin C or E or medications which may impact the results of the ozone challenge (such as, systemic steroids and beta blockers) at least 2 weeks prior to the study and for the duration of the study. Medications not specifically mentioned here may be reviewed by the investigators prior to a subject's inclusion in the study.
* Current and past smokers within 1 year.
* Uncontrolled hypertension (> 150 systolic, > 90 diastolic).
* Subjects who do not understand or speak English
* Subjects unable to perform the moderately active exercise required for the study.
* Subjects with a history of skin allergies to adhesives used in securing heart rate monitor electrodes.
* Unspecified diseases or conditions, which in the judgment of the investigator might influence the responses to the exposures, will be a basis for exclusion.
* Subjects unwilling to stop taking over-the-counter pain medications such as aspirin, Advil, Aleve or other non-steroidal anti-inflammatory medications ("NSAIDS") for 48 hr prior to the exposures and post-exposure visits.
* Subjects with a marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 milliseconds (ms))

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2010-08; Primary Completion 2012-04 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Lung Function Decrement | Immediately post to 24 hr post exposure
  Lung function decrements are typically expressed as changes in FEV1 and FVC. Measurements are made pre-exposure (defined as baseline, immediately post exposure, 1-4 hr post exposure, and 24 hr post exposure (follow up).

SECONDARY OUTCOMES:
Heart rate variability | immediately post to 24 hr post exposure

OTHER OUTCOMES:
plasma cytokine levels | immediately post to 24 hr post exposur
  Inflammation markers such as interleukin 8

CONTACTS AND LOCATIONS:
Overall Officials: Michael Madden, PhD, Principal Investigator — Environmental Protection Agency (EPA)
Locations (1):
- US EPA Human Studies Facility, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Madden MC, Stevens T, Case M, Schmitt M, Diaz-Sanchez D, Bassett M, Montilla TS, Berntsen J, Devlin RB. Diesel exhaust modulates ozone-induced lung function decrements in healthy human volunteers. Part Fibre Toxicol. 2014 Sep 2;11:37. doi: 10.1186/s12989-014-0037-5. PMID 25178924